CLINICAL TRIAL: NCT00145340
Title: The Effect of PPARgamma Stimulation on Glucose Metabolism, Insulin Resistance, Growth Hormone and Cortisol on Women Suffering From Polycystic Ovary Syndrome
Brief Title: Pioglitazone Treatment in Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 032
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome (PCOS); PPARgamma; growth hormone; insulin resistance; pioglitazone; glucose metabolism; microarray
MeSH Terms: conditions — Polycystic Ovary Syndrome; Carotid Intimal Medial Thickness 1; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pioglitazone — 30 Mg/day

SUMMARY:
In this study, the investigators wish to investigate how pioglitazone treatment effects hirsute women. Hirsute women are often overweight and have an increased amount of male sex hormone in their blood. Their blood tests show frequent changes corresponding to the changes seen in diabetic patients.

Pioglitazone is a drug used for increasing the insulin sensitivity in diabetic patients. Previous studies showed that this drug is able to decrease the level of insulin in blood in hirsute women. Moreover, the level of male sex hormones is reduced during this treatment. The drug has only been marketed for few years, and no investigations have been carried out as to the reaction of other hormones, e.g. growth hormone and stress hormone, using this treatment.

This clinical trial includes 30 strongly hirsute women. The patients are randomized to either placebo or an active drug. The treatment period is 16 weeks. The patients included must be healthy and take no medicine possibly changing the results of the study. The patients must take no contraceptive pills or receive any other hormone treatment.

In connection with the investigation, the following will be carried out on all patients: glucose tolerance test, clinical examination, blood tests, measurement of stress hormones and sex hormones, hyperinsulinaemic euglycaemic clamp test, muscle biopsies and bone scan.

This examination programme will be carried out before start of pioglitazone or placebo treatment and again after 16 weeks of treatment. The examinations require 2½ days of hospitalization.

The purpose of the study is to gain more knowledge of the reasons for hirsute women to grow more hair than normal women. The study will show whether pioglitazone treatment can reduce the amount of male sex hormone in blood and how the level of stress hormone and growth hormone is changed when reducing the amount of insulin in blood.

ELIGIBILITY:
Inclusion Criteria:

* Irregular menses, i.e. cyclus length of >36 days
* Premenopausal
* Increased fasting insulin > 50 pmol/l
* Increased free testosterone > 0.035 nmol/l

Exclusion Criteria:

* Age: <18 years
* Contraceptive pill within the past 3 months
* Postmenopausal (increased FSH)
* Known diabetes mellitus, endocrine disease or other disease requiring treatment
* Drug use
* Pregnancy
* Planned pregnancy during the treatment period
* Increased liver parameters

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2002-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Glucose infusion rate (M value) below euglycaemic hyperinsulinaemic clamp (comparing baseline with 4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Glintborg, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Funen, Denmark

REFERENCES:
- [Derived] Glintborg D, Petersen MH, Ravn P, Hermann AP, Andersen M. Comparison of regional fat mass measurement by whole body DXA scans and anthropometric measures to predict insulin resistance in women with polycystic ovary syndrome and controls. Acta Obstet Gynecol Scand. 2016 Nov;95(11):1235-1243. doi: 10.1111/aogs.12964. PMID 27529295
- [Derived] Glintborg D, Hermann AP, Rasmussen LM, Andersen M. Plasma osteoprotegerin is associated with testosterone levels but unaffected by pioglitazone treatment in patients with polycystic ovary syndrome. J Endocrinol Invest. 2013 Jul-Aug;36(7):460-5. doi: 10.3275/8767. Epub 2012 Nov 26. PMID 23211475
- [Derived] Vigerust NF, Bohov P, Bjorndal B, Seifert R, Nygard O, Svardal A, Glintborg D, Berge RK, Gaster M. Free carnitine and acylcarnitines in obese patients with polycystic ovary syndrome and effects of pioglitazone treatment. Fertil Steril. 2012 Dec;98(6):1620-6.e1. doi: 10.1016/j.fertnstert.2012.08.024. Epub 2012 Sep 19. PMID 22999793
- [Derived] Eriksen M, Porneki AD, Skov V, Burns JS, Beck-Nielsen H, Glintborg D, Gaster M. Insulin resistance is not conserved in myotubes established from women with PCOS. PLoS One. 2010 Dec 30;5(12):e14469. doi: 10.1371/journal.pone.0014469. PMID 21209881
- [Derived] Glintborg D, Hojlund K, Andersen NR, Hansen BF, Beck-Nielsen H, Wojtaszewski JF. Impaired insulin activation and dephosphorylation of glycogen synthase in skeletal muscle of women with polycystic ovary syndrome is reversed by pioglitazone treatment. J Clin Endocrinol Metab. 2008 Sep;93(9):3618-26. doi: 10.1210/jc.2008-0760. Epub 2008 Jun 10. PMID 18544618